CLINICAL TRIAL: NCT06539559
Title: Efficacy, Adverse Events and Resistant Mechanism of Eribulin Combined With or Without Bevacizumab for Advanced HER2 Negative Breast Cancer Patients, an Open-label, Randomized, Multi-center PhaseⅡ Clinical Trial.
Brief Title: Efficacy and Resistant Mechanism of Eribulin and Bevacizumab for Advanced HER2 Negative Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wang Jiayu (Other)
Collaborators: Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, Wang Jiayu, Chief Physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CancerIHCAMS-Wjiayu
Record Dates: First submitted 2024-07-28; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Breast Neoplasms; Neoplasm Metastasis; Drug Therapy; Bevacizumab
Keywords: breast cancer; HER2 negative; eribulin; bevacizumab; efficacy; resistant mechanism
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — eribulin; Bevacizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- eribulin+bevacizumab (Experimental): eribulin 1.4 mg/m2 iv d1,8 + bevacizumab 7.5mg/kg ivgtt d1/q21d
  Interventions: Drug: Eribulin; Drug: Bevacizumab
- eribulin (Active Comparator): eribulin 1.4 mg/m2 iv d1,8/q21d
  Interventions: Drug: Eribulin

INTERVENTIONS:
Drug: Eribulin — Based on the results of STUDY301 and STUDY304, eribulin showed outstanding therapeutic effect and tolerable adverse events in patients with metastatic breast cancer
  Other Names: Halaven
Drug: Bevacizumab — Study E2100, AVADO and RIBBON-1 found that in the first-line chemotherapy for advanced breast cancer, the addition of bevacizumab can significantly improve the efficacy of traditional chemotherapy drugs. Study RIBBON-2 and TANIA have confirmed the effectiveness of bevacizumab in the second and third line treatment of advanced HER2 negative breast cancer. Compared with chemotherapy alone, the addition of bevacizumab can prolong the PFS by 0.6 to 2.1 months.
  Other Names: Avastin
  Arms: eribulin+bevacizumab

SUMMARY:
This study is a prospective, multicenter, phase II randomized clinical trial. It is planned to enroll 60 patients with advanced HER2 negative breast cancer, who will be randomly assigned to the experimental group and the control group in a 1:1 ratio. The participants will receive either eribulin combined with bevacizumab or eribulin monotherapy. Every treatment cycle will last for 21 days, with weekly monitoring of blood routine, blood biochemistry and other indicators. Imaging examinations will be conducted every two cycles and the efficacy will be evaluated according to RECIST 1.1 standard. The life quality questionnaire is arranged at baseline and every 3 months after enrollment, and the long-time survival will be followed every 3 months after treatment. The primary endpoint is progression-free survival (PFS), the secondary endpoints are objective response rate (ORR), clinical benefit rate (CBR) and overall survival (OS). The investigators will also focus on the treatment-related adverse events (TRAE) and quality of life (QoL) assessment.

At the same time, this study also aims to explore the resistant mechanisms of anti-angiogenic drugs. The investigators plan to collect peripheral venous blood samples at 3 time points: baseline, during treatment, and end of treatment. All the dynamic samples will be used for transcriptome sequencing to obtain the gene sets. And based on the optimal therapeutic efficacy, all the participants will be divided into response group and non-response group. GO and KEGG enrichment analysis will be subsequently performed between different therapeutic efficacy groups to draw gene interaction networks, identify key action nodes and explain the mechanism of anti-angiogenic drug resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old，and ≤75 years old.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
3. Expected survival period not less than 12 weeks.
4. At least 1 measurable lesion according to RECIST 1.1 standard.
5. previously treated with taxanes and/or anthracycline drugs in any stage of breast cancer.
6. Immunohistochemistry (IHC) and fluorescence in situ hybridization (FISH) validated HER2 negative, including IHC- and IHC 1+/2+ with FISH negative.
7. at least prior 1 line of chemotherapy in the advanced stage.
8. The organ function must meet the following requirements：

(1). Blood Routine

* ANC≥1.5×109/L；
* PLT≥90×109/L；
* Hb≥90 g/L；

  (2). Blood Biochemistry
* TBIL≤1.5×ULN；
* ALT and AST≤2×ULN；ALT和AST≤5×ULN for patients with liver metastasis；
* BUN and Cr≤1.5×ULN and the Creatinine Clearance Rate ≥50 mL/min (Cockcroft-Gault formula calculated)；

  (3). Echocardiogram
* LVEF≥50%；

  (4). electrocardiogram
* The QT interval (QTcF) corrected by Fridericia method less than 450 ms for male and less than 470 ms for female.

  9. Volunteer to join this study, sign informed consent, have good compliance and be willing to cooperate with follow-up.

Exclusion Criteria:

1. There is a third interstitial fluid accumulation that cannot be controlled by drainage or other methods (such as a large amount of hydrothorax and ascites).
2. Symptomatic or uncontrolled brain or meningeal metastases.
3. Patients with only bone or skin metastasis as the assessable lesion.
4. Previously suffered from other malignant tumors.
5. Those who have used Eribulin during the advanced disease stage.
6. Individuals with a known history of allergies to the components of the interventions; History of immunodeficiency, including HIV positive, other acquired or congenital immunodeficiency diseases and a history of organ transplantation.
7. Any heart disease or other conditions evaluated unsuitable by the researcher.
8. Pregnant and lactating female patients, female patients with fertility and positive baseline pregnancy test results, or female patients of reproductive age who are unwilling to take effective contraceptive measures throughout the trial period.
9. According to the investigator's judgment, there are concomitant diseases that seriously endanger the patient's safety or affect the patient's completion of the study (including severe bleeding tendency, history of surgery within 2 weeks, hypertension beyond drug control, serious diabetes, active infection, thyroid disease, etc.).
10. Having a clear history of neurological or mental disorders, including epilepsy or dementia.
11. According to the RECIST 1.1 criteria, researchers determined that patients who received the last anti-tumor regimen before enrollment did not experience disease progression.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | Radiological examinations will be conducted every two cycles: at the end of Cycle 2, 4, 6, 8......(each cycle is 21 days). The PFS will last until disease progression.
  PFS is defined as the time from randomization to the date of confirmed radiological progression or death from any cause.

SECONDARY OUTCOMES:
overall survival (OS) | The long-time survival will be followed every 3 months after the end of treatment.
  OS is defined as the time from randomization to the date of death from any cause and censored at the date of final contact for patients who were still alive.
objective response rate (ORR) | Radiological examinations will be conducted every two cycles: at the end of Cycle 2, 4, 6, 8......(each cycle is 21 days). The efficacy will be evaluated according to RECIST 1.1 standard.
  ORR is defined as the proportion of patients with best response of complete response (CR) and partial response (PR) according to RECIST 1.1 standard.
clinical benefit rate (CBR) | Radiological examinations will be conducted every two cycles and the efficacy will be evaluated according to RECIST 1.1 standard.
  CBR is defined as the proportion of patients with best response of complete response (CR) , partial response (PR) and stable disease (SD) according to RECIST 1.1 standard.

OTHER OUTCOMES:
treatment-related adverse events (TRAE) | Adverse events will be assessed every cycle (each cycle is 21 days) and graded according to the Common Terminology Criteria Adverse Events (CTCAE) version 5 until 1 month after the end of treatment.
  TRAE is defined as the adverse reactions that occur during the use of medication for treatment and are supposed to be related to the intervention drugs.
quality of life (QoL) | The life quality questionnaire is arranged at baseline and every 3 months after enrollment until 6 months after the end of treatment.
  QoL assessment is examined by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire core 30 (EORTC QLQ-C30), of which 30 items were included. Items 1-28 are divided into 4 levels, with ratings ranging from 1 to 4 (the higher score indicates worse life quality). Items 29 and 30 are divided into 7 levels, with ratings ranging from 1 to 7 (the higher score indicates better life quality).

CONTACTS AND LOCATIONS:
Overall Officials: Jiayu Wang, doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (3):
- China (3):
  - Beijing Chaoyang District San Huan Cancer Hospital, Beijing, Beijing Municipality
  - Cancer Hospital of HuanXing ChaoYang District, Beijing, Beijing Municipality
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: After the final analysis of this study on August 2026.

REFERENCES:
- [Background] Hardy-Bessard AC, Brocard F, Clatot F, Lortholary A, You B, Grenier J, Martin-Babau J, Lucas B, Meunier J, Ferrero JM, Savoye AM, Marti A, Despax R, Moullet I, Emile G. First-line bevacizumab and eribulin combination therapy for HER2-negative metastatic breast cancer: Efficacy and safety in the GINECO phase II ESMERALDA study. Breast. 2020 Dec;54:256-263. doi: 10.1016/j.breast.2020.09.011. Epub 2020 Sep 30. PMID 33188992
- [Background] Yuan P, Hu X, Sun T, Li W, Zhang Q, Cui S, Cheng Y, Ouyang Q, Wang X, Chen Z, Hiraiwa M, Saito K, Funasaka S, Xu B. Eribulin mesilate versus vinorelbine in women with locally recurrent or metastatic breast cancer: A randomised clinical trial. Eur J Cancer. 2019 May;112:57-65. doi: 10.1016/j.ejca.2019.02.002. Epub 2019 Mar 29. PMID 30928806
- [Background] Kaufman PA, Awada A, Twelves C, Yelle L, Perez EA, Velikova G, Olivo MS, He Y, Dutcus CE, Cortes J. Phase III open-label randomized study of eribulin mesylate versus capecitabine in patients with locally advanced or metastatic breast cancer previously treated with an anthracycline and a taxane. J Clin Oncol. 2015 Feb 20;33(6):594-601. doi: 10.1200/JCO.2013.52.4892. Epub 2015 Jan 20. PMID 25605862
- [Background] Liu B, Liu L, Ran J, Xie N, Li J, Xiao H, Yang X, Tian C, Wu H, Lu J, Gao J, Hu X, Cao M, Shui Z, Hu ZY, Ouyang Q. A randomized trial of eribulin monotherapy versus eribulin plus anlotinib in patients with locally recurrent or metastatic breast cancer. ESMO Open. 2023 Jun;8(3):101563. doi: 10.1016/j.esmoop.2023.101563. Epub 2023 Jun 6. PMID 37285718
- [Background] von Minckwitz G, Puglisi F, Cortes J, Vrdoljak E, Marschner N, Zielinski C, Villanueva C, Romieu G, Lang I, Ciruelos E, De Laurentiis M, Veyret C, de Ducla S, Freudensprung U, Srock S, Gligorov J. Bevacizumab plus chemotherapy versus chemotherapy alone as second-line treatment for patients with HER2-negative locally recurrent or metastatic breast cancer after first-line treatment with bevacizumab plus chemotherapy (TANIA): an open-label, randomised phase 3 trial. Lancet Oncol. 2014 Oct;15(11):1269-78. doi: 10.1016/S1470-2045(14)70439-5. Epub 2014 Sep 28. PMID 25273342
- [Background] Brufsky AM, Hurvitz S, Perez E, Swamy R, Valero V, O'Neill V, Rugo HS. RIBBON-2: a randomized, double-blind, placebo-controlled, phase III trial evaluating the efficacy and safety of bevacizumab in combination with chemotherapy for second-line treatment of human epidermal growth factor receptor 2-negative metastatic breast cancer. J Clin Oncol. 2011 Nov 10;29(32):4286-93. doi: 10.1200/JCO.2010.34.1255. Epub 2011 Oct 11. PMID 21990397
- [Background] Robert NJ, Dieras V, Glaspy J, Brufsky AM, Bondarenko I, Lipatov ON, Perez EA, Yardley DA, Chan SY, Zhou X, Phan SC, O'Shaughnessy J. RIBBON-1: randomized, double-blind, placebo-controlled, phase III trial of chemotherapy with or without bevacizumab for first-line treatment of human epidermal growth factor receptor 2-negative, locally recurrent or metastatic breast cancer. J Clin Oncol. 2011 Apr 1;29(10):1252-60. doi: 10.1200/JCO.2010.28.0982. Epub 2011 Mar 7. PMID 21383283
- [Result] De Angelis C, Bruzzese D, Bernardo A, Baldini E, Leo L, Fabi A, Gamucci T, De Placido P, Poggio F, Russo S, Forestieri V, Lauria R, De Santo I, Michelotti A, Del Mastro L, De Laurentiis M, Giuliano M, De Placido S, Arpino G. Eribulin in combination with bevacizumab as second-line treatment for HER2-negative metastatic breast cancer progressing after first-line therapy with paclitaxel and bevacizumab: a multicenter, phase II, single arm trial (GIM11-BERGI). ESMO Open. 2021 Apr;6(2):100054. doi: 10.1016/j.esmoop.2021.100054. Epub 2021 Feb 16. PMID 33601296